CLINICAL TRIAL: NCT00838500
Title: Evaluation of the Efficacy of Spa Treatment for Prevention of Leg Ulcers in Advanced Chronic Venous Insufficiency.
Brief Title: THERMES ET VEINES: Spa for Prevention of Leg Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Collaborators: Université Joseph Fourier (Other); Floralis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CUF 1497
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Venous Insufficiency; Leg Ulcer; Varicose Ulcer
Keywords: Venous insufficiency; Leg ulcer; balneology; hydrotherapy; Modified Rutherford score; Euroquol EQ 5d scale; CIVIQ2 scale; Visual analogic Scale; SPA treatment
MeSH Terms: conditions — Venous Insufficiency; Leg Ulcer; Varicose Ulcer

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate SPA treatment (Active Comparator): Immediate spa treatment during 18 days soon after randomization (1 year)
  Interventions: Drug: Immediate spa treatment
- Late SPA treatment (Sham Comparator): Late spa treatment during 18 days soon after 12 months visit (2nd year)
  Interventions: Drug: Late spa treatment

INTERVENTIONS:
Drug: Immediate spa treatment — 1st year, soon after randomization: Spa treatment of 18 days. Spa treatment : the most adapted to the concerned pathology and common to all of spa resorts(walk in a specially pool, whirlpool bath with automatic air and water massages cycles, massaging shower...)
  Arms: Immediate SPA treatment
Drug: Late spa treatment — 2nd year, soon after 12 months visit: Spa treatment of 18 days. Spa treatment : the most adapted to the concerned pathology and common to all of spa resorts(walk in a specially pool, whirlpool bath with automatic air and water massages cycles, massaging shower...)
  Arms: Late SPA treatment

SUMMARY:
The main objective of this study is to test the hypothesis that a 3 week intensive course of spa therapy can reduce the risk of leg ulcers in patients with advanced chronic venous insufficiency (C4a-b and C5 of the CEAP classification) at one year.

DETAILED DESCRIPTION:
Chronic venous insufficiency affects to differing extents half of the French population. The most advanced forms, with skin changes (CEAP clinical classes C4-5-6) affect 5% of the population and are those most often indicated for spa treatment. A venous condition is recognized as justifying spa therapy by 12 spa resorts in France. However, no specific or global benefit has been clearly scientifically shown for such therapy. One methodologically sound study (Carpentier 2009) demonstrated a benefit of spa therapy using a non-clinical intermediate endpoint (severity of skin changes). No study has shown efficacy of spa therapy in the primary and secondary prevention of the major and most common complication of advanced chronic venous insufficiency: leg ulcers.

Vascular hemodynamics and in particular venous return from the lower limbs is subject to the laws of physics. Thus, the roles of the calf muscle venous pump and hydrostatic pressure in venous insufficiency rationalizes the use of balneotherapy techniques in the management of this pathology.

The spa therapy techniques used in the context of venous insufficiency have well-defined physiopathic targets and the hemodynamic and microcirculatory effects of some of them have been demonstrated. The high degree of satisfaction of patients taking the waters annually for venous conditions indirectly testifies to their enhanced well-being. Among venous indications, the prevention of post-thrombotic syndrome is one of the best recognized by the medical profession.Nevertheless, there has been no real validation of this indication with an acceptable methodology that meets the canons of evidence based medicine.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes, more than 18 years old patients with a phlebological indication of spa treatment, with advanced chronic venous insufficiency, class C4a, or b or C5 of CEAP classification (leg ulcers must be healed since 3 months at least)
* Available for a spa treatment during 18 days (immediate or late spa)and a follow-up period of 18 months
* Voluntary to participate to the study,informed consent form signed after appropriate information
* Affiliation to the social security system or equivalent

Exclusion Criteria:

* Pregnancy, parturient or breast feeding
* No psychiatric illness or social situation that would preclude study compliance
* Leg ulcer in progress
* Leg ulcer healed for less than 3 months
* Refusal to consent
* Refusal of spa treatment
* Contra-indication of spa treatment(cancer in progress, psychiatric disorders, immunodeficiency)
* Arteriopathy of lower limb with an Ankle Brachial Pressure Index (ABPI)< 0.7, symptomatic neuropathy, erysipelas within 5 years prior to inclusion
* Surgical or endovascular treatment of the venous disease planned during the first year or during the six months prior to inclusion
* No previous phlebological spa treatment within 6 months prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of a leg ulcer within the year following the inclusion. The ulcer will be classified C5 of CEAP (healed ulcer) or C6 (non healed ulcer)at the follow up visit. | 1 year

SECONDARY OUTCOMES:
Healing time of the leg ulcers within the first year | 12 months
Quality of life: Euroqol EQ 5D, CIVIQ2 Scale | Inclusion - 6 months - 12 months- 18 months
Aggravation level defined as at least 20% increase of the modified Rutherford score and mean comparison of this score at 1 year | Inclusion - 12 months - 18 months
Visual analog scale for leg symptoms | Monthly (until 18 months)
Evaluation of the costs involved by the venous insufficiency at 1 year (treatments, physical treatments, hospitalization) | Inclusion - 6, 12 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick PC CARPENTIER, Professor, Principal Investigator — Grenoble Hospital - France
Locations (13):
- France (13):
  - Cabinet médical, Albertville
  - Cabinet médical, Angoulême
  - Cabinet médical, Bagnoles-de-l'Orne
  - Cabinet médical, Barbotan-les-Thermes
  - Cabinet médical, Bayonne
  - Cabinet médical, Belfort
  - Hopital thermal, Dax
  - University Hospital Grenoble, Grenoble
  - Cabinet médical, Montluçon
  - Cabinet médical, Montpellier
  - Cabinet médical, Pau
  - Cabinet médical, Rochefort
  - Cabinet médical, Tarbes

REFERENCES:
- [Background] Carpentier PH, Maricq HR, Biro C, Poncot-Makinen CO, Franco A. Prevalence, risk factors, and clinical patterns of chronic venous disorders of lower limbs: a population-based study in France. J Vasc Surg. 2004 Oct;40(4):650-9. doi: 10.1016/j.jvs.2004.07.025. PMID 15472591
- [Background] Carpentier PH, Satger B. Randomized trial of balneotherapy associated with patient education in patients with advanced chronic venous insufficiency. J Vasc Surg. 2009 Jan;49(1):163-70. doi: 10.1016/j.jvs.2008.07.075. Epub 2008 Oct 1. PMID 18829219
- [Background] Ernst E, Saradeth T, Resch KL. A single blind randomized, controlled trial of hydrotherapy for varicose veins. Vasa. 1991;20(2):147-52. PMID 1877335
- [Background] Eklof B, Rutherford RB, Bergan JJ, Carpentier PH, Gloviczki P, Kistner RL, Meissner MH, Moneta GL, Myers K, Padberg FT, Perrin M, Ruckley CV, Smith PC, Wakefield TW; American Venous Forum International Ad Hoc Committee for Revision of the CEAP Classification. Revision of the CEAP classification for chronic venous disorders: consensus statement. J Vasc Surg. 2004 Dec;40(6):1248-52. doi: 10.1016/j.jvs.2004.09.027. PMID 15622385
- [Background] Rutherford RB, Padberg FT Jr, Comerota AJ, Kistner RL, Meissner MH, Moneta GL. Venous severity scoring: An adjunct to venous outcome assessment. J Vasc Surg. 2000 Jun;31(6):1307-12. doi: 10.1067/mva.2000.107094. PMID 10842165
- [Background] Launois R, Reboul-Marty J, Henry B. Construction and validation of a quality of life questionnaire in chronic lower limb venous insufficiency (CIVIQ). Qual Life Res. 1996 Dec;5(6):539-54. doi: 10.1007/BF00439228. PMID 8993100
- [Background] Constant F, Collin JF, Guillemin F, Boulange M. Effectiveness of spa therapy in chronic low back pain: a randomized clinical trial. J Rheumatol. 1995 Jul;22(7):1315-20. PMID 7562765
- [Background] Labropoulos N, Leon LR Jr. Duplex evaluation of venous insufficiency. Semin Vasc Surg. 2005 Mar;18(1):5-9. doi: 10.1053/j.semvascsurg.2004.12.002. PMID 15791546
- [Background] Prandoni P, Lensing AW, Prins MH, Frulla M, Marchiori A, Bernardi E, Tormene D, Mosena L, Pagnan A, Girolami A. Below-knee elastic compression stockings to prevent the post-thrombotic syndrome: a randomized, controlled trial. Ann Intern Med. 2004 Aug 17;141(4):249-56. doi: 10.7326/0003-4819-141-4-200408170-00004. PMID 15313740
- [Derived] Carpentier PH, Blaise S, Satger B, Genty C, Rolland C, Roques C, Bosson JL. A multicenter randomized controlled trial evaluating balneotherapy in patients with advanced chronic venous insufficiency. J Vasc Surg. 2014 Feb;59(2):447-454.e1. doi: 10.1016/j.jvs.2013.08.002. Epub 2013 Oct 15. PMID 24135621
- See also: e_crf test website (username: THERMES99 - Passwor:thermestst) — https://www.clininfohosting.com/specif/THERMES/